CLINICAL TRIAL: NCT06994026
Title: Feasibility Study of a Relapse Investigation Questionnaire Administered by an MS Care Coordinator Nurse in Patients With Multiple Sclerosis
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier de Gonesse (Other)
Responsible Party: Sponsor
Other Study IDs: 0062_NEUROLOGIE_TIPO
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Multiple Sclerosis; Disease Management; Feasibility Studies
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate a questionnaire used by a specialized nurse to help manage relapses in people with multiple sclerosis (MS). The questionnaire is completed during a phone call when the patient reports new or worsening symptoms. It helps the nurse decide whether further tests or treatments are needed, based on a protocol developed with a neurologist. The goal is to improve how quickly and effectively patients receive care during a relapse. The study will include 10 adult patients with active forms of MS over a two-month period.

ELIGIBILITY:
Inclusion Criteria:

* Patients followed by Dr. Manchon for Relapsing-Remitting Multiple Sclerosis or active Secondary Progressive Multiple Sclerosis
* Adult patients (aged 18 or older)
* Patients who have provided informed consent for participation in the local task-sharing protocol

Exclusion Criteria:

* Pregnant women
* Minors (under 18 years old)
* Patients with known renal failure
* Patients who have not provided or are unable to provide consent for the local task-sharing protocol

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The participants will be selected from adult patients with Multiple Sclerosis (MS) who are under the care of Dr. Manchon at a single neurology center. Specifically, the population includes individuals diagnosed with either Relapsing-Remitting MS or active Secondary Progressive MS. All participants must have provided informed consent to be included in a local task-sharing protocol that allows a specialized nurse (IDEC) to conduct initial evaluations during suspected relapses. This population reflects patients who are actively monitored for MS and may experience acute neurological symptoms requiring timely assessment and intervention.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of the relapse investigation questionnaire completed by the MS care coordinator nurse (IDEC) in guiding the patient's care pathway during a suspected relapse, according to the local task-sharing protocol. | June 2025 - August 2025

CONTACTS AND LOCATIONS:
Locations (1):
- France, Gonesse, France, France